CLINICAL TRIAL: NCT05510609
Title: Three-dimensional Ultrasonography: Accuracy in Thyroid Volume Measurement.
Brief Title: Three-dimensional Ultrasonography Thyroid Volume Measurement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Klara Bay Rask, Stud.Med., Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-22011900
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Thyroid; Thyroid Cancer; Thyroid Diseases; Graves Disease; Thyroid Goiter; Thyroid Adenoma
Keywords: Ultrasound; Ultrasonography; Volumetry; Thyroid Gland; Three Dimensional; 3D
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms; Graves Disease; Goiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thyroidectomy (Other): Patients set for total thyroidectomy incl. functional total thyroidectomies.
  Interventions: Device: BK 5000 Ultrasound Machine

INTERVENTIONS:
Device: BK 5000 Ultrasound Machine — Both 2D and 3D ultrasound is being used. 3D using optical tracking.

SUMMARY:
The purpose of this clinical trial is to investigate the accuracy of applying three-dimensional ultrasound on thyroid gland patients when determining a gland volume.

The method will be compared to conventional b-mode ultrasound where three axis measurements (length, width, and depth) are evaluated in the ellipsoid model.

The three dimensional (3D) method is utilizing optical tracking connected to the ultrasound image to form cross-sectional imaging. Patients enrolled in the study are set for complete thyroidectomies enabling a true volume of the gland by water displacement after excision.

The aim is to find if this 3D method is more accurate in volume estimation than the ellipsoid model.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to Rigshospitalet to undergo a complete thyroidectomy including patients with previous hemithyroidectomy
* Adults, 18 or older.
* Ability to give written informed consent

Exclusion Criteria:

* Thyroid glands that are too enlarged causing visualization/measurement impairment with ultrasonography.
* Thyroid cancer with preoperative suspected extracapsular spread.
* Thyroids or lymph nodes that need frozen section examination.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Thyroid volume | 1 hour
  Obtaining thyroid volume with 2D ultrasound (length x Width x depth*(Pi/6)) and 3D ultrasound with optical tracking and comparing the respective methods with a reference volume. Water displacement being gold standard for reference volume.

SECONDARY OUTCOMES:
Shrinkage in gland after excision | 30 minutes
  Looking af the change in volume invivo vs exvivo w. 2D and 3D ultrasound
Interobserver variability | 2 hours
  Variation in volume estimation when delineating ultrasound images.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capital, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reinartz P, Sabri O, Zimny M, Nowak B, Cremerius U, Setani K, Bull U. Thyroid volume measurement in patients prior to radioiodine therapy: comparison between three-dimensional magnetic resonance imaging and ultrasonography. Thyroid. 2002 Aug;12(8):713-7. doi: 10.1089/105072502760258695. PMID 12225640
- [Result] van Isselt JW, de Klerk JM, van Rijk PP, van Gils AP, Polman LJ, Kamphuis C, Meijer R, Beekman FJ. Comparison of methods for thyroid volume estimation in patients with Graves' disease. Eur J Nucl Med Mol Imaging. 2003 Apr;30(4):525-31. doi: 10.1007/s00259-002-1101-1. Epub 2003 Jan 23. PMID 12541136
- [Result] Brunn J, Block U, Ruf G, Bos I, Kunze WP, Scriba PC. [Volumetric analysis of thyroid lobes by real-time ultrasound (author's transl)]. Dtsch Med Wochenschr. 1981 Oct 9;106(41):1338-40. doi: 10.1055/s-2008-1070506. German. PMID 7274082
- [Result] Schlogl S, Werner E, Lassmann M, Terekhova J, Muffert S, Seybold S, Reiners C. The use of three-dimensional ultrasound for thyroid volumetry. Thyroid. 2001 Jun;11(6):569-74. doi: 10.1089/105072501750302877. PMID 11442004
- [Result] Freesmeyer M, Knichel L, Kuehnel C, Winkens T. Stitching of sensor-navigated 3D ultrasound datasets for the determination of large thyroid volumes - a phantom study. Med Ultrason. 2018 Dec 8;20(4):480-486. doi: 10.11152/mu-1687. PMID 30534656
- [Result] Freesmeyer M, Wiegand S, Schierz JH, Winkens T, Licht K. Multimodal evaluation of 2-D and 3-D ultrasound, computed tomography and magnetic resonance imaging in measurements of the thyroid volume using universally applicable cross-sectional imaging software: a phantom study. Ultrasound Med Biol. 2014 Jul;40(7):1453-62. doi: 10.1016/j.ultrasmedbio.2014.02.013. Epub 2014 Apr 24. PMID 24768486
- [Result] Seifert P, Winkens T, Knichel L, Kuhnel C, Freesmeyer M. Stitching of 3D ultrasound datasets for the determination of large thyroid volumes - phantom study part II: mechanically-swept probes. Med Ultrason. 2019 Nov 24;21(4):389-398. doi: 10.11152/mu-2006. PMID 31765446
- [Result] Boers T, Braak SJ, Versluis M, Manohar S. Matrix 3D ultrasound-assisted thyroid nodule volume estimation and radiofrequency ablation: a phantom study. Eur Radiol Exp. 2021 Jul 29;5(1):31. doi: 10.1186/s41747-021-00230-4. PMID 34322765
- [Result] Lyshchik A, Drozd V, Reiners C. Accuracy of three-dimensional ultrasound for thyroid volume measurement in children and adolescents. Thyroid. 2004 Feb;14(2):113-20. doi: 10.1089/105072504322880346. PMID 15068625
- [Result] Malago R, D'Onofrio M, Ferdeghini M, Mantovani W, Colato C, Brazzarola P, Motton M, Mucelli RP. Thyroid volumetric quantification: comparative evaluation between conventional and volumetric ultrasonography. J Ultrasound Med. 2008 Dec;27(12):1727-33. doi: 10.7863/jum.2008.27.12.1727. PMID 19022998
- [Result] Andermann P, Schlogl S, Mader U, Luster M, Lassmann M, Reiners C. Intra- and interobserver variability of thyroid volume measurements in healthy adults by 2D versus 3D ultrasound. Nuklearmedizin. 2007;46(1):1-7. PMID 17299648
- [Result] Jang M, Kim SM, Lyou CY, Choi BS, Choi SI, Kim JH. Differentiating benign from malignant thyroid nodules: comparison of 2- and 3- dimensional sonography. J Ultrasound Med. 2012 Feb;31(2):197-204. doi: 10.7863/jum.2012.31.2.197. PMID 22298862
- [Result] Kim SC, Kim JH, Choi SH, Yun TJ, Wi JY, Kim SA, Sun HY, Ryoo I, Park SW, Sohn CH. Off-site evaluation of three-dimensional ultrasound for the diagnosis of thyroid nodules: comparison with two-dimensional ultrasound. Eur Radiol. 2016 Oct;26(10):3353-60. doi: 10.1007/s00330-015-4193-2. Epub 2016 Jan 22. PMID 26795614
- [Result] Ng E, Chen T, Lam R, Sin D, Ying M. Three-dimensional ultrasound measurement of thyroid volume in asymptomatic male Chinese. Ultrasound Med Biol. 2004 Nov;30(11):1427-33. doi: 10.1016/j.ultrasmedbio.2004.09.004. PMID 15588952
- [Result] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Result] AIUM practice guideline for the performance of ultrasound examinations of the head and neck. J Ultrasound Med. 2014 Feb;33(2):366-82. doi: 10.7863/ultra.33.2.366. No abstract available. PMID 24449746
- [Result] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Derived] Rask KB, Makouei F, Wessman MHJ, Kristensen TT, Todsen T. Thyroid Volume Measurement With AI-Assisted Freehand 3D Ultrasound Compared to 2D Ultrasound-A Clinical Trial. Head Neck. 2026 Jan;48(1):64-70. doi: 10.1002/hed.28267. Epub 2025 Aug 8. PMID 40778496